CLINICAL TRIAL: NCT02720939
Title: ASD-specific Induced Pluripotent Stem Cells for Disease Modeling
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201507086RINA
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood will be collected in the INSEPACK Disposable Vacuum Venous Blood Specimen collection Tube (Green Tube with li-Heparin) and each tube will contain 5-10ml of blood from ASD probands and healthy controls.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ASD group: ASD patients who met the diagnostic criteria of either autistic disorder or Asperger's disorder defined by the DSM-IV criteria
- TD group: Typically development controls without lifetime diagnosis with ASD or any psychiatric disorders

SUMMARY:
Specific Aims:

1. To generate induced-pluripotent stem cells (iPSCs) from peripheral blood mononuclear cells (PBMCs) isolated from whole blood of ASD probands and healthy controls.
2. To derive neural progenitor cells (NPCs) and neurons from iPSCs of ASD probands and healthy controls and compare differences between patients and healthy controls to investigate the cellular phenotype of ASD and uncover the pathophysiology of the disease.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) is a common, lifelong impairing childhood-onset neurodevelopmental disorder with clinical and genetic heterogeneity. The etiology of ASD is complicated and remains largely unknown. Evidences indicate the high heritability (54-77%) in ASD, and researchers also found copy number variations (CNVs) play an important role in the etiology of ASD. However, due to the ethical issue, researchers haven't had an appropriate platform to investigate the copy number change effect to date. In the following study, researchers are going to derive ASD-specific induced pluripotent stem cells and neurons for disease modeling.

10 ASD patients and 10 healthy controls will be included in the present study and iPSCs and neurons will be generated from their PBMCs. Electrophysiological recording and analysis of neuronal morphology will be conducted to reveal the cellular phenotype of ASD after comparing differences between patients and healthy controls.

The study will provide a platform to reveal the etiology of genetic basis and molecular mechanism of ASD. The cellular phenotype of ASD will be revealed by comparing differences between patients and healthy controls. The findings from this work are expected to contribute to the basic and clinical research on ASD.

ELIGIBILITY:
Inclusion Criteria:

* ASD group: Subjects who met the diagnostic criteria of either autistic disorder or Asperger's disorder defined by the DSM-IV criteria.

Exclusion Criteria:

* TD group: Subjects with any current or lifetime DSM-IV psychiatric disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample will consist of 10 ASD patients and 10 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
iPSC derivation and characterization | 12 weeks
  To generate induced-pluripotent stem cells (iPSCs) from peripheral blood mononuclear cells (PBMCs) isolated from whole blood of ASD probands and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan